CLINICAL TRIAL: NCT03854721
Title: Phase I Safety and Tolerability of Intravesical VAX014 for Instillation in Subjects With Non-Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: A Phase 1 Study of Intravesical VAX014 for Instillation in Subjects With Non-Muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxiion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX0116
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Urothelial Carcinoma of the Urinary Bladder
Keywords: Non-Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VAX014 (Experimental): Intravesical VAX014 (dose: 3.33x10^10 - 9.0x10^11 recombinant bacterial minicells (rBMCs)), given once per week for Weeks 1-6
  Interventions: Drug: VAX014

INTERVENTIONS:
Drug: VAX014 — Solution for intravesical infusion, 3.33x10^10 rBMCs per vial

SUMMARY:
The purpose of this research study is to evaluate the safety, tolerability and activity of VAX014 for Instillation (VAX014) in patients with low-grade Non-Muscle Invasive Bladder Cancer (NMIBC). VAX014 is a targeted oncolytic agent designed to kill tumor cells following instillation into the urinary bladder.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of VAX014 using a 3+3 dose escalation design to determine a maximum tolerated dose (MTD) followed by a dose expansion at the Recommended Phase 2 Dose (RP2D). Both phases of the study will use a Window of Opportunity study design where patients with a single, low-grade Ta lesion will receive VAX014 via a urinary catheter into the bladder, weekly for 6 weeks prior to undergoing Transurethral Resection of Bladder Tumor (TURBT) to assess antitumor activity against the mapped lesion.

Patients enrolled in this study must have low-grade (Ta) Non-Muscle Invasive Bladder Cancer. However, eligible patients may have up to 5 low-grade Ta lesions at screening, and all but a single mapped lesion will be resected prior to receiving VAX014. The mapped lesion is assessed for anti-tumor activity.

VAX014 is a formulation of recombinant bacterial minicells which is designed to selectively target two NMIBC-associated integrin heterodimers to de-stabilize tumor cell membranes, with the result being tumor cell lysis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent
2. Age 18 or more years
3. Pathologically confirmed low-grade Ta urothelial carcinoma (UC) of the urinary bladder
4. NMIBC with one solitary measurable tumor at the start of study, measuring ≥ 5 mm and ≤ 15 mm in greatest diameter (up to 4 additional low-grade Ta lesions, each measuring no more than 15 mm may be removed at screening provided a single lesion remains)
5. Treatment-naïve or failed one previous regimen of intravesical therapy (BCG or chemotherapy)
6. If recurrent disease, then more than 6 months from prior resection, more than 3 months from completion of last intravesical therapy with BCG, and more than 6 weeks from completion of last therapeutic intravesical therapy with chemotherapy
7. If previously treated, recovered from prior treatment-related toxicity to ≤ Grade 1
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 116
9. Absolute neutrophil count (ANC) ≥ 1,500/mm3
10. Platelet count ≥ 100,000/mm3
11. Total bilirubin ≤ 1.5 x upper limit of normal (ULN), or ≤ 3 x ULN in subjects with Gilberts disease
12. Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 30 mL/min
13. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x ULN
14. Willingness to participate in collection of pharmacokinetic samples
15. Women of childbearing potential must have a negative serum pregnancy test.
16. All subjects of childbearing potential must be willing to use effective contraception while on treatment and for 3 months after the last dose of VAX014

Exclusion Criteria:

1. Additional papillary disease at screening (in addition to the solitary low-grade Ta lesion detailed in the inclusion criteria) that

   1. Consist of 6 or more lesions
   2. Consists of any lesion with a maximal diameter of greater than 15 mm
2. Confirmed or suspected perforated bladder
3. History of difficult catheterization that in the opinion of the investigator will prevent administration of VAX014
4. Presence or history of any high-grade urothelial cancer (including CIS) or high-grade urine cytology
5. Intravesical chemo-or biological therapy within 6 months of first administration of VAX014
6. UC of the ureters or urethra
7. History of interstitial cystitis
8. History of radiation to the pelvis
9. History of vesicoureteral reflux or an indwelling urinary stent
10. Other known active cancer(s) likely to require treatment or interfere with study objectives over the next two (2) years
11. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
12. Known HIV, Hepatitis B, or Hepatitis C infection
13. Significant cardiovascular risk (e.g., coronary stenting within 8 weeks, myocardial infarction within 6 months)
14. Major surgery other than diagnostic surgery within 4 weeks of first administration of VAX014
15. Pregnant or currently breast-feeding
16. Psychiatric illness/social situations that would interfere with compliance with study requirements
17. Presence of any sessile appearing tumor suspected of being invasive or high-grade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of VAX014 | up to 28 days
  The MTD will be defined as the dose level at which at most one of six patients experiences a dose limiting toxicity (DLT) after 28 days of treatment have occurred, with the next higher dose having at least 2/3 or 2/6 patients experiencing a DLT
Incidence of Treatment-Emergence Adverse Events (Safety and Tolerability) | Through study completion, an average of 20 weeks
  Toxicities will be assessed in each subject by tracking the occurrence of graded Adverse Events (AEs). AEs will be graded according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) v5.0

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of intravesical VAX014 | up to 5 weeks
  The RP2D will be determined following the determination of the MTD and an overall assessment of safety as determined by the Safety Committee
Peak Plasma Concentration (Cmax) | Day 1
  The peak plasma concentration (Cmax) will be measured as part of pharmacokinetic (PK) testing. In the event early analysis determines that VAX014 is not detectable in whole blood, PK sampling and analysis will be suspended.
Trough Plasma Concentration (Cmin) | Day 1
  The trough plasma concentration (Cmin) will be measured as part of pharmacokinetic (PK) testing. In the event early analysis determines that VAX014 is not detectable in whole blood, PK sampling and analysis will be suspended.
Time to Peak Plasma Concentration (Tmax) | Day 1
  The time to peak plasma concentration (Tmax) will be measured as part of pharmacokinetic (PK) testing. In the event early analysis determines that VAX014 is not detectable in whole blood, PK sampling and analysis will be suspended.
Volume and Distribution (Vd) | Day 1
  The volume and distribution (Vd) will be measured as part of pharmacokinetic (PK) testing. In the event early analysis determines that VAX014 is not detectable in whole blood, PK sampling and analysis will be suspended.
Half Life (t[1/2]) | Day 1
  The half life (t[1/2]) will be measured as part of pharmacokinetic (PK) testing. In the event early analysis determines that VAX014 is not detectable in whole blood, PK sampling and analysis will be suspended.
Area Under Curve (AUC) | Day 1
  The area under the plasma concentration versus time curve (AUC) will be measured as part of pharmacokinetic (PK) testing. In the event early analysis determines that VAX014 is not detectable in whole blood, PK sampling and analysis will be suspended.
Clearance (Cl) | Day 1
  The clearance (Cl) will be measured as part of pharmacokinetic (PK) testing. In the event early analysis determines that VAX014 is not detectable in whole blood, PK sampling and analysis will be suspended.
Overall Response Rate | Up to 20 weeks
  Response rate will be evaluated for low-grade Ta lesions. Lesions will be assessed with cystoscopy and change in tumor size will be recorded.
Anti-Drug Antibodies (Immunogenicity) | Up to 20 weeks
  The presence or absence of anti-drug antibodies (ADA) in serum will be assessed by assay.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Urology Center of Colorado, Denver, Colorado
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - New Jersey Urology, LLC., Edison, New Jersey
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No